CLINICAL TRIAL: NCT06993545
Title: Impact of Promoting Physical Exercise on Migraine - a Video-based Randomized Clinical Trial
Brief Title: Educational Video Program to Promote Physical Activity and Reduce Migraine Frequency in Adults With Migraine
Acronym: PA-MIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 393/2023
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Migraine Disorders; Exercise; Health Education; Audiovisual Aids; Surveys and Questionnaires
Keywords: Migraine disorders; exercise; health education; audiovisual aids; surveys and questionnaires
MeSH Terms: conditions — Migraine Disorders; Motor Activity; Health Education

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group received usual care provided by their healthcare professionals, with no additional educational materials or interventions related to physical activity. This group did not receive the video-based educational program. Throughout the study, preventive and acute treatments were maintained according to standard clinical practice. Participants completed the same assessments as the intervention group at baseline and follow-up, including questionnaires on migraine impact, frequency, medication use, and physical activity levels.
- Intervention group (Experimental): The intervention consisted of a series of seven short, pre-recorded educational videos delivered over a 3-month period. The videos focused on the benefits of regular physical activity for individuals with migraine and included practical strategies to increase daily activity levels. The content was evidence-based, developed with input from healthcare professionals, and tailored to migraine management. Participants received access to one video approximately every two weeks via email or online platform. The videos aimed to improve awareness, motivation, and self-efficacy regarding physical activity without prescribing a specific exercise program. No direct interaction with healthcare providers occurred during the intervention period.
  Interventions: Behavioral: Video-based educational program on physical activity for migraine management

INTERVENTIONS:
Behavioral: Video-based educational program on physical activity for migraine management — The intervention consisted of a series of seven short, pre-recorded educational videos delivered over a 3-month period. The videos focused on the benefits of regular physical activity for individuals with migraine and included practical strategies to increase daily activity levels. The content was evidence-based, developed with input from healthcare professionals, and tailored to migraine management. Participants received access to one video approximately every two weeks via email or online platform. The videos aimed to improve awareness, motivation, and self-efficacy regarding physical activity without prescribing a specific exercise program. No direct interaction with healthcare providers occurred during the intervention period.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn if an educational video program can help reduce migraine frequency and improve migraine-related outcomes in adults with migraine. The main questions it aims to answer are:

* Does the video-based intervention reduce the number of monthly migraine episodes?
* Does it reduce the use of acute migraine medication?
* Does it increase the physical activity levels?

Researchers will compare participants who watch educational videos about physical activity with participants who receive usual care, to see if the intervention has additional benefits.

Participants will:

* Be randomly assigned to one of two groups: intervention or control
* The intervention group will watch seven short educational videos over a period of 3 months
* All participants will complete questionnaires before and after the intervention period to assess migraine impact, frequency, medication use, and physical activity levels

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosis of episodic or chronic migraine confirmed by a neurologist, based on the 3rd edition of the International Classification of Headache Disorders (ICHD-3)
* Willing and able to participate in the study

Exclusion Criteria:

* Inability to read or understand the study materials
* Inability or unwillingness to collaborate with study procedures
* Refusal to participate
* Diagnosis of other primary headache disorders (except for medication overuse headache)
* Presence of substance use disorders
* Presence of chronic medical conditions that limit physical activity (e.g., rheumatic diseases, systemic inflammatory conditions, neoplastic diseases)
* Presence of severe psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Change in Headache Impact Test (HIT-6) score from baseline to 6-month follow-up | HIT-6 scores were collected at baseline (T0) and at 6-month follow-up (T6), corresponding to three months after the completion of the video-based intervention.
  The Headache Impact Test (HIT-6) is a validated questionnaire used to assess the impact of headaches on a person's ability to function in daily life. It includes six questions covering domains such as pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. Each item is scored on a scale, and the total score ranges from 36 to 78, with higher scores indicating greater impact of headaches. In this study, HIT-6 was used as the primary outcome measure to evaluate the effect of the video-based educational intervention on migraine-related disability. Scores were collected at baseline and again six months later, three months after the intervention period ended, to assess any changes in the perceived impact of migraine on participants' lives.

SECONDARY OUTCOMES:
Change in physical activity indices from baseline to 6-month follow-up in the intervention group | Assessed at baseline (T0) and 6-month follow-up (T6), corresponding to three months after the intervention period.
  Three physical activity indices (PAI) were used to evaluate changes in participants' activity levels: job-related PAI, housework, house maintenance, and caring for family-related PAI, and recreation, sport, and leisure time-related PAI. These indices are derived from validated self-report questionnaires and reflect both the intensity and frequency of physical activity in different contexts. This outcome aimed to assess whether the video-based educational intervention led to meaningful behavioral changes regarding physical activity. Measurements were taken at baseline and again at 6-month follow-up, corresponding to three months after the completion of the video series.
Change in monthly migraine frequency from baseline to 6-month follow-up in the intervention group | Assessed at baseline and at 6-month follow-up (T6), i.e., three months post-intervention.
  Migraine frequency was measured as the number of self-reported migraine days per month. This secondary outcome aimed to evaluate whether the educational video program contributed to a reduction in the frequency of migraine attacks. Participants recorded their migraine occurrences in headache diaries, and data were collected at baseline and at the 6-month follow-up to compare the frequency before and after the intervention.
Change in monthly frequency of acute medication use from baseline to 6-month follow-up in the intervention group | Reported monthly and compared between baseline and 6-month follow-up, which occurred three months after the intervention.
  This outcome measures how often participants used acute medication (e.g., analgesics or triptans) to treat migraine attacks each month. The goal was to determine whether the video-based educational program reduced the need for acute migraine medication. Participants kept monthly medication logs, and frequency data were collected at baseline and again at the 6-month follow-up to evaluate the impact of the intervention.
Patient Global Impression of Change (PGIC) score at 6-month follow-up in the intervention group | Assessed only at the 6-month follow-up (T6), three months after completion of the intervention.
  At the 6-month follow-up, participants' perceived overall change in their migraine condition was assessed using an adapted version of the Patient Global Impression of Change (PGIC) scale. This version was translated and culturally adapted to Portuguese and asked participants to rate how their condition had changed since the beginning of the study. Response options ranged from "no changes (or worsening of the condition)" to "much better." The PGIC is a validated, subjective measure commonly used in chronic condition trials to evaluate patients' impressions of treatment effectiveness. This outcome aimed to capture participants' global self-assessment of improvement or deterioration after the educational video intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade Local de Saúde de São João, E.P.E., Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided